CLINICAL TRIAL: NCT00899691
Title: Detection and Quantification of Changes in Levels of Protein Expression and Phosphorylation Status Using Human Hair Samples
Brief Title: Study of Hair Samples From Patients With Cancer
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: 040138; 04-C-0138; CDR0000363803
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

INTERVENTIONS:
Genetic: protein expression analysis

SUMMARY:
RATIONALE: Studying samples of hair in the laboratory from patients with cancer may help doctors identify biomarkers related to cancer and predict how well patients will respond to treatment.

PURPOSE: This laboratory study is looking at hair samples from patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether layered membrane technology can quantitatively measure the expression, activity, and localization of cell growth control and signaling proteins in hair samples from patients with cancer.
* Correlate changes in protein expression with expected changes based on planned therapy in these patients.

OUTLINE: This is a pilot, multicenter study.

Hair samples are obtained from patients at baseline and at the end of study. The samples are assayed for proteins and phosphorylation status using layered membrane technology. Proteins analyzed may include vascular endothelial growth factor receptor (VEGFR), Erk1/2, Akt, epidermal growth factor receptor (EGFR), and c-KIT.

PROJECTED ACCRUAL: A total of 190 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of malignancy
* Undergoing treatment at the National Cancer Institute's Clinical Center
* Must have scalp hair

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2005-03; Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Obtain data on the detection and quantification of changes in levels of protein expression and phosphorylation status using human hair samples at baseline and after completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Steven K. Libutti, MD, Principal Investigator — NCI - Surgery Branch